CLINICAL TRIAL: NCT01320839
Title: Effects of an Ankle-Foot Orthosis on Gait While Performing an Attention Demanding Task in People With Poststroke Hemiplegia
Brief Title: Effects of an Ankle-Foot Orthosis on Gait While Performing an Attention Demanding Task
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Kim Parker, Rehabilitation Engineer, Nova Scotia Health Authority
Other Study IDs: CDHA-RS/2011-004
Record Dates: First submitted 2011-02-23; First posted 2011-03-23 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Stroke; Gait, Hemiplegic
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stroke: People who have had a stroke and have an ankle-foot orthosis.

SUMMARY:
We hypothesize that: (1) gait stability will be increased when wearing an ankle-foot orthosis (plastic brace supporting the foot and ankle); (2) an attention demanding task will decrease gait stability and (3) the improvement in gait stability due to ankle-foot orthosis use will be greater during an attention demanding task.

DETAILED DESCRIPTION:
A quasi-experimental, randomized 2 x 2 factorial within subjects study with the factor of walking condition (2 levels, walking with and without ankle-foot orthotic device) and attention condition (2 levels, walking with and without attention task).

ELIGIBILITY:
Inclusion Criteria:

* be over the age of 18;
* have the presence of hemiplegia after stroke;
* be wearing an ankle-foot orthosis for at least 6 weeks;
* be able to walk independently and comfortably for a minimum distance of 12 m with or without assistive aids (AFOs, canes and walkers);
* be able to read and understand English, follow verbal instructions and provide verbal answers to questions;
* be able to reach criterion on the attention task (described below)
* be competent to give informed consent as determined by clinical team and noted in the health chart

Exclusion Criteria:

* have history of balance deficits not related to stroke;
* be at high risk of falling during the study;
* suffer from severe aphasia or dementia as determined by health chart and/or initial cognitive screening using the Montreal Cognitive Assessment (MoCA) test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have had a hemiplegic stroke and have an ankle-foot orthosis.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Velocity | up to one week
  walking velocity

SECONDARY OUTCOMES:
trunk acceleration | up to one week
  trunk acceleration during walking
Step length variability | up to one week
  variability of right and left step length during walking
The Berg Balance Scale | up to one week
  Functional balance measured using the Berg Balance Scale short form.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Parker, M.A.Sc., Principal Investigator — CDHA
Locations (1):
- Capital Health, Halifax, Nova Scotia, Canada